CLINICAL TRIAL: NCT01812876
Title: A Registry Study on Shenqifuzheng（a Chinese Medicine Injection）Used in Hospitals in China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy Director, China Academy of Chinese Medical Sciences
Other Study IDs: 2009ZX09502-030-01
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Gastric Carcinoma; Carcinoma of the Lungs
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: None Retained — Eligibility criteria Patients who will use Shenqifuzheng injection in selected hospitals.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study was advocated by Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences in December 2012.

It was funded by China major scientific and technological specialized project for 'significant new formulation of new drugs'.

The purpose of this study is to make a cohort event monitoring to see whether and how Shenqifuzheng injection in hospital results in adverse events or adverse drug reactions.

DETAILED DESCRIPTION:
It is very common that Chinese Medicine Injection used in hospitals in mainland China. However safety problems rose in recent years. There could be many uncertain factors influence Chinese Medicine Injection in clinical practice.

Safety surveillance on Chinese Medicine injection is an important problem that needs to be sorted out through large sample observational study.

A registry study for Shenqifuzheng injection safety surveillance with 30000 patients will be conducted from Jan.2013 to Dec.2014.

Eligibility criteria Patients who will use Shenqifuzheng injection in selected hospitals

ELIGIBILITY:
Inclusion Criteria:

- Patients using Shenqifuzheng injection from 2013 to 2014

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An anticipated sample size was caculated in this study, about 30000 Patients using Shenqifuzheng injection from 2013 to 2014 in more than 30 hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events; incidence of Shenqifuzheng'ADRs and identify factors that contributed to the occurrence of the adverse reaction | to assess Shenqifuzheng's 'adverse event' and 'drug adverse reaction' during patients' hospital stay, administration information of Shenqifuzheng will be registered every day. The registry procedure will last 3 years only for patients using Shenqifuzheng
  All patients will be measured and assessed at the time Shenqifuzheng is administered to them until they discharge. Patients using Shenqifuzheng will be registered on a registration form including disease background, Shenqifuzheng's administration, and extraction information from hospital information system. An adverse event or drug adverse reaction form also will be used to describe any doubted symptoms or signs from patients. A judgment will be made by doctors directly and a further analysis will be conducted by researchers to decide those potential side effects of Shenqifuzheng

CONTACTS AND LOCATIONS:
Overall Officials: Xie M Yan, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences